CLINICAL TRIAL: NCT02239861
Title: Tumor Associated Antigen (TAA)-Specific Cytotoxic T-Lymphocytes Administered to Patients With Solid Tumors
Brief Title: TAA-Specific CTLS for Solid Tumors (TACTASOM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other); Solving Kids' Cancer (Other); Pierce Phillips Charity (Unknown)
Responsible Party: Principal Investigator, Sarah Whittle, Assistant Professor, Pediatric Hematology/Oncology, Center for Cell and Gene Therapy, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-35425, TACTASOM
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Rhabdomyosarcoma
Keywords: Rhabdomyosarcoma; cytotoxic T lymphocytes
MeSH Terms: conditions — Rhabdomyosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAA-Specific CTLs (Experimental): 4 different dosing schedules will be evaluated. 2 to 4 patients will be evaluated on each dosing schedule. The first 2 patients on each dose level will be staggered by 4 weeks (which starts when the first infusion is given, Day 0). No subjects between the ages of 2-18 will be enrolled to a dose level on this protocol, until an adult has been enrolled to and treated on that dose level on one of the protocols being conducted under this same IND. Each patient will receive 2 injections at the same dose,14 days apart: The expected volume of infusion will be 1 to 10 cc.
  Dose Level One:
  Day 0 and 14: 5 x 10^6 cells/m^2
  Dose Level Two:
  Day 0 and 14: 1 x 10^7 cells/m^2
  Dose Level Three:
  Day 0 and 14: 2 x 10^7 cells/m^2
  Dose Level Four:
  Day 0 and 14: 4 x 10^7 cells/m^2
  Interventions: Biological: TAA-Specific CTLs

INTERVENTIONS:
Biological: TAA-Specific CTLs — Patients may be pre-medicated with Benadryl up to 1 mg/kg IV (max 50 mg) and Tylenol 10 mg/kg po (max 650 mg).
  Cell Administration: Tumor-specific T cells will be given by intravenous injection over 1-10 minutes through either a peripheral or a central line.
  Patients with stable disease or better will receive up to 6 further doses of CTLs, as long as they continue to show disease stabilization or improvement by RECIST criteria at their 8 week or subsequent evaluations. Each dose will consist of the same number as their second injection or less (if there is not enough product available for the subject's original dose).
  Patients will not be able to receive additional doses until the initial safety profile is completed at 6 weeks following the second infusion.
  Other Names: Tumor Associated Antigen-Specific Cytotoxic T-Lymphocytes

SUMMARY:
This is a clinical trial for patients with a solid tumor which has come back, or may come back, or has not gone away after treatment, including the standard treatment we know for these diseases. This is a study using special immune system cells called tumor-associated antigen (TAA)-specific cytotoxic T lymphocytes, a new experimental therapy.

The proteins that the investigators are targeting in this study are called tumor-associated antigens (TAAs). These are cell proteins that are specific to the cancer cell, so they either do not show or show up in low quantities on normal human cells. In this study, the investigators target five common TAAs called NY-ESO-1, MAGEA4, PRAME, Survivin and SSX. On a different study, patients have been treated and so far this treatment has shown to be safe.

The investigators now want to try this treatment in patients with solid tumors.

This protocol is designed as a Phase I dose-escalation study.

DETAILED DESCRIPTION:
Blood will be collected from the patient and TAA-specific CTLs will be made.

The cells will be injected by IV into the patient over 1 - 10 minutes. The patient may be pre-treated with acetaminophen (Tylenol) and diphenhydramine (Benadryl). Acetaminophen (Tylenol) and diphenhydramine (Benadryl) are given to prevent a possible allergic reaction to the T cell infusion. Initially, two doses of T cells will be given two weeks apart. The patient's disease will be assessed pre-infusion and then 6 weeks after the second infusion. If after the second infusion, there is a reduction in size of the patient's tumor or if the tumor remains stable on CT or MRI scan as assessed by a radiologist, the patient can receive up to six (6) additional doses of the T cells at monthly intervals. All of the treatments will be given by the Center for Cell and Gene Therapy at Houston Methodist Hospital or Texas Children's Hospital.

In between the first and second T cell infusions, and for 6 weeks after the last infusion, the investigators ask that the patient not receive any other anti-cancer treatments, such as radiation therapy or chemotherapy, except PD1/PDL1 inhibitors as clinically indicated. If the patient does receive any other therapies in-between the first and second infusion of T cells, they will be taken off treatment and will not be able to receive the second infusion of T cells.

This is a dose escalation study. This means that at the beginning, patients will be started on the lowest dose (1 of 4 different levels) of T cells. Once that dose schedule proves safe, the next group of patients will be started at a higher dose. This process will continue until all 4 dose levels are studied. If the side effects are too severe, the dose will be lowered or the T cell injections will be stopped.

MEDICAL TESTS BEFORE TREATMENT:

Before being treated, patients will receive a series of standard medical tests:

* Physical exam.
* Blood tests to measure blood cells, kidney and liver function.
* Measurements of the patient's tumor by routine imaging studies. The investigators will use the imaging study that was previously performed to follow the patient's tumor: Computer Tomogram (CT), Magnetic Resonance Imaging (MRI), or Positron Emission Tomography (PET).
* Pregnancy test if the patient is a female who can have children.

MEDICAL TEST AFTER TREATMENT:

Patients will receive standard medical test after infusion:

* Patients will receive standard medical test after infusion:
* Blood tests to measure blood cells, kidney and liver function.
* Imaging study 6 weeks after the 2nd CTL infusion.

To learn more about the way the T cells are working in the patient's body, an extra 20-40 mL (4-8 teaspoons) of blood will be taken before each infusion, and at Weeks 1, 2, 4 and 6. Afterwards, blood will be collected at 3, 6, 9 and 12 months after the last infusion. The investigators will use this blood to see how long the T cells last, and to look at the immune response to the patient's response to cancer. Patients will then be contacted once a year for up to 4 additional years (total of 5 years follow-up) to evaluate their disease response long-term.

Study Duration: The patient's active participation in this study will last for approximately one (1) year. If the patient receives additional doses of the TAA-CTLs as described above, then the patient's active participation will last until one (1) year after his/her last dose. We will then contact the patient once a year for up to 4 additional years (total of 5 years follow-up) in order to evaluate his/her disease response long-term.

ELIGIBILITY:
THIS PROTOCOL IS CURRENTLY NOT RECRUITING ADULTS.

Procurement Inclusion Criteria:

1. Any patient regardless of sex with a solid tumor expressing any of the following antigens (PRAME, SSX2, MAGEA4, NY-ESO1-1 and/or Survivin) with:

   1. Active disease after first line therapy;
   2. Refractory disease;
   3. As adjuvant therapy for high risk disease (high risk disease is a disease that has a >50% risk of progression within 5 years)
2. Patients with life expectancy at least 6 weeks.
3. Age greater than or equal to 2 and less than or equal to 80 years old.
4. Hgb >8.0
5. Informed Consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.

Procurement Exclusion Criteria:

1. Diagnosis of primary CNS tumor.
2. Patients with severe intercurrent infection.
3. Patients with active HIV infection at time of procurement (can be pending at the time of blood draw).
4. Patients in remission who are enrolled on another study where time to progression or disease-free survival is a primary endpoint.

Treatment Inclusion Criteria:

1. Any patient regardless of sex with a solid tumor expressing any of the following antigens (PRAME, SSX2, MAGEA4, NY-ESO1-1 and/or Survivin) with:

   1. Active disease after first line therapy;
   2. Refractory disease;
   3. As adjuvant therapy for high risk disease (high risk disease is a disease that has a >50% risk of progression within 5 years)
2. Patients with life expectancy at least 6 weeks.
3. Age greater than or equal to 2 and less than or equal to 80 years old.
4. Pulse oximetry of >95% on room air in patients who previously received radiation therapy.
5. Patients with a Karnofsky/Lansky score of greater than or equal to 50.
6. Patients with bilirubin less than or equal to 2x upper limit of normal, AST less than or equal to 3x upper limit of normal, and Hgb >8.0
7. Patients with a creatinine less than or equal to 2x upper limit of normal for age.
8. Patients should have been off other investigational therapy for one month prior to entry in this study.
9. Patients should have been off conventional therapy for at least 1 week prior to entry in this study. PD1/PDL1 inhibitors will be allowed if medically indicated.
10. Informed Consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.
11. Due to unknown effects of this therapy on a fetus, pregnant women are excluded from this research. The male partner should use a condom Females of child-bearing potential must be willing to utilize one of the more effective birth control methods during the study unless female has had a hysterectomy or tubal ligation.

Treatment Exclusion Criteria:

1. Diagnosis of primary CNS tumor.
2. Patients with severe intercurrent infection.
3. Patients receiving systemic corticosteroids (patients off steroids for at least 48 hours are eligible).
4. Pregnant or breastfeeding
5. HIV positive.
6. Patients in remission who are enrolled on another study where time to progression or disease-free survival is a primary endpoint.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose-limiting toxicity. | 8 weeks
  The Phase I dose escalation trial is designed for the primary goal of evaluating the safety and feasibility of administering TAA-CTLs to patients with solid tumors.

SECONDARY OUTCOMES:
Number of patients with a disease response to the CTLs. | 8 weeks
  The Phase I dose escalation trial is designed for the primary goal of evaluating the safety and feasibility of administering TAA-CTLs to patients with solid tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Leen, PhD, Principal Investigator — Baylor College of Medicine; Cliona Rooney, PhD, Principal Investigator — Baylor College of Medicine; Helen Heslop, MD, Principal Investigator — Baylor College of Medicine; Sarah Whittle, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas